CLINICAL TRIAL: NCT06747312
Title: A Single Center, Randomized Controlled, Open Label Trial to Explore the Regulatory Effect of Belimumab on Antibody Titers in Primary Antiphospholipid Syndrome Patients Carrying Medium to High Titers of Antiphospholipid Antibodies
Brief Title: Effect of Belimumab on Antibody Titers in Primary APS Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024136
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-07

CONDITIONS: Antiphospholipid Syndrome (APS)
Keywords: Belimumab; Antiphospholipid Syndrome (APS); Antiphospholipid Antibodies
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: SOC+Belimumab arm (Experimental): Belimumab 10mg/kg once a month as an add-on treatment regimen. SOC treatment includes aspirin and/or vitamin K antagonists (VKA) and/or low molecular weight heparin.
  Interventions: Drug: Belimumab+SOC; Drug: SOC
- Experimental: SOC arm (Active Comparator): SOC treatment includes aspirin and/or vitamin K antagonists (VKA) and/or low molecular weight heparin.
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: Belimumab+SOC — 10mg/kg once a month for 18 months
  Arms: Experimental: SOC+Belimumab arm
Drug: SOC — SOC treatment includes aspirin and/or vitamin K antagonists (VKA) and/or low molecular weight heparin.

SUMMARY:
The purpose of this study is to evaluate the regulatory effect of Belimumab on the antiphospholipid antibody (aPL) as well as to observe related past and new clinical events in primary antiphospholipid syndrome patients.

DETAILED DESCRIPTION:
This is a single center, randomized controlled trial in Ruijin Hospital. The enrolled patients will be randomized in a 1: 1 ratio to receive either SOC+Belimumab or SOC treatment. Belimumab is administered intravenously at a dose of 10mg/kg once a month for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Positive for high-titer antiphospholipid antibodies according to the criteria of the "EULAR Guidelines for the Treatment of Antiphospholipid Syndrome in Adults" published in 2019.
* Stable APS regimen according to EULAR recommendations for antiphospholipid syndrome.
* Female patients who are not pregnant, breastfeeding, of childbearing potential, or not using contraception.

Exclusion Criteria:

* Patients with a history of malignant tumor in the past 5 years, except for basal cell carcinoma or squamous cell carcinoma of skin or cervical carcinoma in situ treated locally, and there is no evidence of metastasis within 3 years;
* Patients with a history of primary immunodeficiency;
* Serious lack of IgG (IgG level < 400 mg/dL);
* IgA deficiency (IgA level < 10 mg/dL);
* Patients with a current history of infection;
* Patients with a current history of drug or alcohol abuse or dependence, or have a history of drug or alcohol abuse or dependence within 365 days before day 0;
* HIV test is historically positive or HIV screening is positive;
* Hepatitis status;
* Patients with a history of allergic reaction caused by injection of contrast agent, human or mouse protein or monoclonal antibody;
* Patients with other abnormal laboratory values with clinical significance;
* If women with reproductive potential (WCBP) are included, please refer to the following special instructions;
* Patients with concurrent major medical or mental illnesss;
* Patients with diseases of liver, kidney, heart and other important organs,blood and Endocrine system;
* Patients who have been vaccinated with live vaccine in the last month;
* Patients who have participated in any clinical trial within 28 days before the initial screening and/or within 5 times of the half-life of the study compound (whichever is longer);
* Patients who use B-cell targeted therapy drugs within one year, such as rituximab or epratuzumab;
* Patients who use tumor necrosis factor inhibitor and interleukin receptor blocker within one year;
* Patients who use Intravenous gamma globulin (IVIG) and prednisone ≥100mg/d for more than 14 days within one year or plasma exchange;
* Patients with active infection (such as herpes zoster, HIV infection, active tuberculosis, etc.) during the screening period;
* Patients with depression or suicidal thoughts;
* Other conditions that the investigator considers would make the candidate unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The level of antiphospholipid antibody titers | 18 months

SECONDARY OUTCOMES:
New thrombotic event | 18 months
  Any new thrombotic event during Belimumab treatment
Effects of Belimumab on the genotype, phenotype, and functional heterogeneity of T and B cells | 18 months
  Application of single-cell RNA sequencing technology (scRNAseq)

OTHER OUTCOMES:
The incidence and severity of adverse events | 18 months
  Number and intensity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China